CLINICAL TRIAL: NCT06426017
Title: Impact of FTO Gene Variation on Body Composition, Lipid Profile, Insulin Resistance, Advanced Glycation End-Products and Ghrelin Levels in Response to Hypocaloric, Protein Rich-Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Bibi Hajira, Assistant Professor, Khyber Medical University Peshawar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMU/IBMS/IRBE/2023/1209-20
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Obesity; Insulin Resistance; Dyslipidemias; Advance Glycation; Inflammation
Keywords: Satiety; Food Intake; High protein diet; Obesity; FTO rs9939609; Ghrelin; Carboxymethyl lysine; Interleukin-6
MeSH Terms: conditions — Obesity; Insulin Resistance; Dyslipidemias; Inflammation

STUDY DESIGN:
Intervention Model Description: It will be a quasi-experimental study, where 110 individuals with obesity will be allocated into three allele groups i.e. TT, AT and AA based on minor allele frequency. Each participant in the study will go through intervention of high protein, low calorie diet for four weeks.
  BMI, waist to hip ratio, body composition, lipid profile, fasting glucose level, insulin resistance, advanced glycation end-products will measure at the start and end of the study while hunger hormone will be measured at the start, mid and end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- High Protein Low Calorie Diet (Experimental): 3 meals/day consumed by the participants with daily caloric intake of 800 kcal. 40-60% of the total calories added from both animal and plant proteins. 30% of the total calories added from fats. 20% of the total calories added from carbohydrates.
  Interventions: Other: High Protein Low Calorie Dietary Intervention

INTERVENTIONS:
Other: High Protein Low Calorie Dietary Intervention — High Protein Diet: Diet consisting of 40-60% total energy from proteins, <20% total energy from carbohydrates and <30% total energy from fats.

SUMMARY:
Obesity is a widespread disease that basically develops from unhealthy lifestyle and genetics. The Fat-mass and obesity associated (FTO) gene affects appetite and energy intake of the body, thus elevating fat mass and body weight. The single nucleotide polymorphism (SNP) rs9939609 of the FTO gene is a common variant in different ethnic groups, and its A allele is associated with increased body mass and waist circumference. Hence, the carriers of rs9939609 SNP are prone to weight gain if a healthy diet and lifestyle are not maintained. Similarly, high levels of serum cholesterol and triglycerides, while low levels of high-density lipoproteins are observed in carriers of rs9939609 AA genotype. For individuals having FTO rs9939609 A allele, consumption of hypocaloric diets (1500 kcal/day) consisting of high protein foods up to 25-30% of total daily energy intake might help reduce body weight. However, weight loss tends to vary in individuals after consuming the same diet under similar environmental conditions, so it is important to know the effect of different genotypes that might cause this variation. The study aimed to genotype overweight and obese adults for FTO rs9939609 polymorphism and to determine the effect of this polymorphism on body weight, BMI, waist and hip circumferences, lipid profile, insulin sensitivity, ghrelin levels, inflammatory markers and advanced glycation end-products in these individuals after consumption of a hypocaloric, high-protein diet for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1Overweight (BMI ≥ 25kg/m2) and obese (BMI ≥ 30kg/m2) individuals.
* Both genders.
* Age 18-50 years.

Exclusion Criteria:

* Children, pregnant and lactating women
* Individuals taking medication for weight loss or undergoing any other weight loss dietary intervention.
* Individuals having lost more than 5 pounds in the past three-month period.
* Patients with any psychiatric disorders, heart, liver, kidney disease, diabetes or abnormal thyroid function.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Body Composition | Day 0 and day 29
  Body composition will be measured using Bioimpedance scale which will include percent body fatness, muscle mass, total body water, bone mass and body protein status.
Lipid Profile | Day 0 and day 29
  Lipid profile will include concentration of total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides in blood and measured in mg/dl.
Waist Circumference | Day 0 and day 29
  Waist circumference will measured in cm using a non-stretchable tape.
Hip Circumference | Day 0 and day 29
  Hip circumference will measured in cm using a non-stretchable tape.
HOMA-IR | Day 0 and day 29
  HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) will be reported in pmol/L.
Serum Carboxymethyl lysine levels (CML) | Day 0 and day 29
  Sreum concentration of Carboxymethyl lysine (CML) will be used an advanced glycation endproduct (AGE) marker and expressed in ng/mL.
Serum Interleukinin-6 (IL-6) | Day 0 and day 29
  Serum Interleukinin-6 (IL-6) will be used as marker of inflammation pg/mL.
Serum Hunger Hormone- Ghrelin | Day 1(Fasting and postprandial), Day 7(Fasting and postprandial) and Day 28(Fasting and postprandial).
  Serum Hunger Hormone- Ghrelin will be used to asses satiety related sensation and expressed as pmol/l.
Body Mass Index (BMI) | Day 0 and day 29
  Body weight will be measured in Kg. Height will be measure in cm. Weight and height will be used to calculate body mass index (BMI) to report in Kg/m^2
Waist-to-Hip Ratio (WHR) | Day 0 and Day 29
  Waist and Hip Circumference will be measured in cm. These two measures will be used to calculate waist-to-hip ratio (WHR) as waist measurement divided by hip measurement (W⁄H).

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Khyber Medical University, Peshawar, KPK
  - Trial Room Institute of Basic Medical Sciences, Peshawar, KPK

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rexrode KM, Carey VJ, Hennekens CH, Walters EE, Colditz GA, Stampfer MJ, Willett WC, Manson JE. Abdominal adiposity and coronary heart disease in women. JAMA. 1998 Dec 2;280(21):1843-8. doi: 10.1001/jama.280.21.1843. PMID 9846779
- [Background] McMillan DC, Sattar N, McArdle CS. ABC of obesity. Obesity and cancer. BMJ. 2006 Nov 25;333(7578):1109-11. doi: 10.1136/bmj.39042.565035.BE1. No abstract available. PMID 17124223
- [Background] Karra E, O'Daly OG, Choudhury AI, Yousseif A, Millership S, Neary MT, Scott WR, Chandarana K, Manning S, Hess ME, Iwakura H, Akamizu T, Millet Q, Gelegen C, Drew ME, Rahman S, Emmanuel JJ, Williams SC, Ruther UU, Bruning JC, Withers DJ, Zelaya FO, Batterham RL. A link between FTO, ghrelin, and impaired brain food-cue responsivity. J Clin Invest. 2013 Aug;123(8):3539-51. doi: 10.1172/JCI44403. Epub 2013 Jul 15. PMID 23867619
- [Background] Zou ZC, -J Mao L, Shi YY, Chen JH, Wang LS, Cai W. Effect of exercise combined with dietary intervention on obese children and adolescents associated with the FTO rs9939609 polymorphism. Eur Rev Med Pharmacol Sci. 2015 Dec;19(23):4569-75. PMID 26698254